CLINICAL TRIAL: NCT01463085
Title: A Randomized, Controlled, Trial to Assess the Effects of Low-fat Dairy Intake on Endothelial Function and Blood Pressure in Subjects With Pre-hypertension or Stage 1 Hypertension
Brief Title: Clinical Trial to Assess the Effects of Low-fat Dairy on Systolic Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dairy Research Institute (Other)
Collaborators: BioFortis (Other); Provident Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRV-11022
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control foods (Placebo Comparator): 3 servings per day of control foods
  Interventions: Other: Low-fat dairy
- Low-fat dairy (Experimental): 3 servings per day of low-fat dairy products
  Interventions: Other: Low-fat dairy

INTERVENTIONS:
Other: Low-fat dairy — Dietary Intervention of 3 servings per day of low-fat dairy

SUMMARY:
The purpose of this study is to determine if increased consumption of low-fat dairy can reduce blood pressure and improve endothelial function in men and women with pre or stage-1 hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female or male, 20-69 years of age, inclusive.
* Subject has a BMI of 18.5 to 39.9 kg/m2, inclusive.
* Subject has resting blood pressure measurements meeting the criteria for pre-hypertension (SBP = 120 to 139 mm Hg and/or DBP = 80 to 89 mm Hg) or stage 1 hypertension (SBP = 140 to 159 mm Hg or DBP = 90 to 99 mm Hg)
* Subject reports history of consuming, on average, ≤2 servings/d of dairy foods as part of their normal diet
* Subject is willing to consume ≤1 serving/d of dairy foods (other than the study products provided) during each treatment phase.
* Subject is willing to maintain a stable body weight and habitual diet and physical activity patterns throughout the trial, with the exception of specific study instructions related to study product intake, alcohol intake, and physical activity.

Exclusion Criteria:

* Subject has known coronary heart disease (CHD) or a CHD risk equivalent
* Subject has a history of any major trauma or major surgical event
* Subject has digital deformities that would prevent EndoPAT measurements.
* Subject has used medications known to alter body weight
* Subject has used medications or dietary supplements that, in the opinion of the Investigator, have strong potential to influence blood pressure or endothelial function
* Subject has extreme dietary habits (e.g., Atkins diet, very high protein/low carbohydrate).

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 5 weeks
  Seated, resting blood pressure and heart rate will be measured by an automated blood pressure measurement device.

SECONDARY OUTCOMES:
Vascular function | 5 weeks
  Subjects will be fasted overnight and endothelial function will be determined using the EndoPAT System according to the manufacturer's instructions. The measurements will occur in the index fingers of both hands, simultaneously and will be taken with subjects in a sitting position while in a quiet, thermo- neutral room.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — Biofortis - Provident Clinical Research
Locations (1):
- Biofortis - Provident Clinical Research, Glen Ellyn, Illinois, United States